CLINICAL TRIAL: NCT06237725
Title: The Effect of Abdominal Massage on Gastrointestinal System Functions in Patients Nutrition Enterally With Continuous and Bolus Infusion.
Brief Title: Abdominal Massage in Enteral Nutrition Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Assoc. Prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MassageGIS
Record Dates: First submitted 2023-11-25; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Enteral Nutrition; Gastrointestinal System--Abnormalities
Keywords: Enteral Nutrition; Continuous and Bolus Infusion; Abdominal Massage; Gastrointestinal System Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nutrition of Continuous (Experimental): Experimental: Intervention Group to Nutrition of Continuous
  Interventions: Other: Nutrition of Continuous
- Control Group Nutrition of Continuous (No Intervention): Control Group to Nutrition of Continuous
- Nutrition of Bolus (Experimental): Experimental: Intervention Group to Nutrition of Bolus
  Interventions: Other: Nutrition of Bolus
- Control Group Nutrition of Bolus (No Intervention): Control Group to Nutrition of Bolus

INTERVENTIONS:
Other: Nutrition of Continuous — The researcher will perform gastric residual volume (GRV) measurements with a syringe, abdominal circumference measurements, and distension assessments daily before starting enteral nutrition from the first day of initiation. They will also record vomiting/defecation frequency. Massage will be applied for 15 minutes. The same criteria will be measured and recorded. The application and measurements will be conducted twice a day for 10 consecutive days.
  Arms: Nutrition of Continuous
Other: Nutrition of Bolus — The researcher will perform gastric residual volume (GRV) measurements with a syringe, abdominal circumference measurements, and distension assessments daily before starting enteral nutrition from the first day of initiation. They will also record vomiting/defecation frequency. Massage will be applied for 15 minutes. The same criteria will be measured and recorded. The application and measurements will be conducted twice a day for 10 consecutive days.
  Arms: Nutrition of Bolus

SUMMARY:
Complications related to the gastrointestinal system may arise in patients receiving enteral nutrition through continuous and bolus infusion. These complications include constipation, diarrhea, nausea, vomiting, abdominal distension, increased gastric residual volume, and abdominal pain. The aim of this study is to determine the impact of abdominal massage applied to patients receiving enteral nutrition through continuous or bolus infusion on gastrointestinal system functions. For this purpose, 164 patients meeting the inclusion criteria will be randomized, and four groups will be defined. Half will constitute the experimental group, and the others will form the control group. In our study, the effects of massage on symptom control will be evaluated by comparing symptoms in patients receiving both forms of nutrition. Thus, the evaluation and control of medical conditions (symptoms) such as constipation, diarrhea, vomiting, increased abdominal distension, and increased gastric residual volume are targeted.

ELIGIBILITY:
Inclusion Criteria:

* Patients in intensive care
* Those aged 18 and above
* Patients being fed through a nasogastric tube
* Patients on the first day of enteral nutrition
* Patients without wounds in the abdominal region
* Those who have not undergone abdominal surgery in the last 6 months
* Patients not receiving radiotherapy/chemotherapy
* Patients without a diagnosis of bowel obstruction
* Patients without diarrhea and constipation
* Patients with a Glasgow Coma Scale (GKS) > 3
* Those with an APACHE II score > 16
* Patients not taking prokinetic agents
* Patients not taking laxative medications
* Patients without any contraindications for abdominal massage (to be determined in consultation with the primary physician)

Exclusion Criteria:

* Patients for whom enteral nutrition is discontinued during the study
* Patients with interrupted enteral nutrition
* Patients who have started prokinetic agents
* The study will be terminated for patients who have started laxative medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Gastric residual volume | 7 days
  GRV measurement will be made 30 minutes after stopping feeding. It will be evaluated before and after application.
Abdominal Distension | 7 days
  Abdominal distension will be evaluated 30 minutes after stopping feeding. The palpation method will be used. Additionally, the abdominal circumference will be measured with a tape measure. It will be evaluated before and after application.
Bowel sounds | 7 days
  Bowel sounds should be evaluated 30 minutes after stopping feeding. Bowel sounds are listened to with a stethoscope for one minute. It will be evaluated before and after the application.

SECONDARY OUTCOMES:
Defecation patterns | 7 days
  measure defecation frequency and nature
Vomiting | 7 days
  How many times the patient vomited during the day is recorded

REFERENCES:
- [Background] Uysal N, Eser I, Akpinar H. The effect of abdominal massage on gastric residual volume: a randomized controlled trial. Gastroenterol Nurs. 2012 Mar-Apr;35(2):117-23. doi: 10.1097/SGA.0b013e31824c235a. PMID 22472671
- [Background] Wang X, Sun J, Li Z, Luo H, Zhao M, Li Z, Li Q. Impact of abdominal massage on enteral nutrition complications in adult critically ill patients: A systematic review and meta-analysis. Complement Ther Med. 2022 Mar;64:102796. doi: 10.1016/j.ctim.2021.102796. Epub 2021 Dec 10. PMID 34902566
- [Background] Dehghan M, Malakoutikhah A, Ghaedi Heidari F, Zakeri MA. The Effect of Abdominal Massage on Gastrointestinal Functions: a Systematic Review. Complement Ther Med. 2020 Nov;54:102553. doi: 10.1016/j.ctim.2020.102553. Epub 2020 Sep 12. PMID 33183670
- [Background] Cetinkaya O, Ovayolu O, Ovayolu N. The Effect of Abdominal Massage on Enteral Complications in Geriatric Patients. SAGE Open Nurs. 2020 Oct 13;6:2377960820963772. doi: 10.1177/2377960820963772. eCollection 2020 Jan-Dec. PMID 35155761
- [Background] Zhang W, Zhou W, Kong Y, Li Q, Huang X, Zhao B, Su H, Chen S, Shen X, Qiu Z. The effect of abdominal massage on enteral nutrition tolerance in patients on mechanical ventilation: A Randomized Controlled Study. Intensive Crit Care Nurs. 2023 Apr;75:103371. doi: 10.1016/j.iccn.2022.103371. Epub 2022 Dec 15. PMID 36528462